CLINICAL TRIAL: NCT05262426
Title: Optimizing an mHealth Intervention to Improve Uptake and Adherence of the HIV Pre-exposure Prophylaxis (PrEP) in Vulnerable Adolescents and Emerging Adults
Brief Title: Developing mHealth to Promote PrEP Use Among Thai Young Vulnerable Adolescents and Emerging Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Wayne State University (Other); Institute of HIV Research and Innovation Foundation, Thailand (Other)
Responsible Party: Principal Investigator, Bo Wang, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: H00023527; 1R21HD107988-01 (NIH)
Record Dates: First submitted 2022-02-07; First posted 2022-03-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pre-Exposure Prophylaxis
Keywords: Pre-exposure Prophylaxis (PrEP); HIV Prevention; mHealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard PrEP Counseling, MES-PrEP and Enhanced YaCool (Experimental): Participants in this arm will receive standard PrEP counseling, followed by two mHealth interventions (MES-PrEP and Enhanced YaCool) to improve PrEP uptake and support PrEP adherence.
  Interventions: Behavioral: Behavioral: Motivational Enhancement System for PrEP Uptake and Adherence (MES-PrEP); Behavioral: Enhanced YaCool; Behavioral: Standard PrEP Counseling
- Standard PrEP Counseling and MES-PrEP (Experimental): Participants in this arm will receive standard PrEP counseling, followed by one mHealth intervention (MES-PrEP) to improve PrEP uptake and support PrEP adherence.
  Interventions: Behavioral: Behavioral: Motivational Enhancement System for PrEP Uptake and Adherence (MES-PrEP); Behavioral: Standard PrEP Counseling
- Standard PrEP Counseling and Enhanced YaCool (Experimental): Participants in this arm will receive standard PrEP counseling, followed by one mHealth intervention (Enhanced YaCool) to improve PrEP uptake and support PrEP adherence.
  Interventions: Behavioral: Enhanced YaCool; Behavioral: Standard PrEP Counseling
- Standard PrEP Counseling (Active Comparator): Participants in this arm will receive the standard PrEP counseling.
  Interventions: Behavioral: Standard PrEP Counseling

INTERVENTIONS:
Behavioral: Behavioral: Motivational Enhancement System for PrEP Uptake and Adherence (MES-PrEP) — MES-PrEP is a two-session computer-delivered intervention based on IMB model. The intervention is tailored based on the person's ratings of perceived importance and confidence of initiating PrEP and sustaining adherence to PrEP. Participants are routed to different intervention content based on their assessment of their importance and confidence. Youth are provided with feedback on scores on the knowledge assessment followed by information about protective effect that can result from improved PrEP adherence. Finally, participants are asked to set a goal: obtain PrEP prescription, optimal adherence, practice steps, or thinking about it more, and they form plans for overcoming barriers. In the second session, branches are based on whether the youth felt they met the goal, partially met the goal, or did not meet the goal. Sessions of MES-PrEP will occur at baseline and month 1.
  Arms: Standard PrEP Counseling and MES-PrEP; Standard PrEP Counseling, MES-PrEP and Enhanced YaCool
Behavioral: Enhanced YaCool — Enhanced YaCool is mobile application developed to support transgender women self-management of their gender and sexual health, including PrEP use. YaCool is a passcode-protected app that allows users to personalized text messaged reminders to take PrEP and/or clinic appointments, record PrEP adherence and sexual activity, and track lab tests. The application is set up to provide personalized recommendations for PrEP regimen, confirmed by clinic healthcare staff. Participants will be asked to download Enhanced YaCool to support PrEP use and gender/sexual health self-management between MES-PrEP sessions for 30 days, and thereafter until the end of Month 12 (if desired).
  Arms: Standard PrEP Counseling and Enhanced YaCool; Standard PrEP Counseling, MES-PrEP and Enhanced YaCool
Behavioral: Standard PrEP Counseling — All participants will received one-on-one, face to face counseling from lay providers at baseline, months 1, 3, 6, 9 and 12. Standard PrEP counseling includes sexual and behavioral risk assessment for HIV/STIs and risk reduction. For those not on PrEP, the sessions will focus on risk perception, awareness of PrEP/post-exposure prophylaxis (PEP) and facilitators and barriers of accessing PrEP. For those on PrEP, the sessions will focus on adherence. Standard counseling sessions will be nonjudgmental, non-discriminatory and client-centered.

SUMMARY:
The main aim of this study is to develop technology-based interventions to improve HIV pre-exposure prophylaxis (PrEP) uptake and adherence among Thai young transgender women.

DETAILED DESCRIPTION:
Motivational Enhancement System for Adherence (MESA) is a computer-based motivation invention, based on the Information-Motivation-Behavioral Skills (IMB) model and Motivational Interviewing (MI) principles, used to promote adherence among HIV-positive youth initiating antiretroviral treatment. In this study, the team will adapt and develop MESA to focus on PrEP uptake and adherence, which will be called Motivational Enhancement System for PrEP Uptake and Adherence (MES-PrEP). YaCool is a mobile application developed to support transgender women self-management of gender and sexual health, including PrEP use.

In Aim 1, the investigators will begin with needs assessment to evaluate intervention efficacy by exploring the barriers and facilitators of PrEP uptake and adherence through in-depth interviews with transgender women and community health workers. The two interventions will be developed and refined based upon the inputs from transgender women through focus group discussion and community advisory board.

In Aim 2, the investigators will conduct a Multiphase Optimization Strategy (MOST) design-based trial to evaluate the feasibility, acceptability, and preliminary efficacy of MES-PrEP and Enhanced YaCool and to determine whether MES-PrEP works better when combined with Enhanced YaCool to improve PrEP use. Eligible transgender women will be randomized to one of the four experimental conditions, and followed for 12 months with assessments at baseline, month 1, 3, 6, 9 and 12.

ELIGIBILITY:
Aim 1:

Transgender women participants

Inclusion Criteria:

* Age 16-29 years old
* Male sex at birth
* Self-identifies as woman or transgender women or culturally identifies with the female spectrum
* Confirmed HIV-negative status
* Self-reported recent history of condomless sex in the past 6 months
* Able to understand, read and speak Thai
* Either having not started PrEP (Group 1: PrEP naive), currently on PrEP but not adherent to PrEP (taking ≤3 pills/week) in the past month (Group 2: PrEP users) or currently on PrEP with good adherence (Group 3: PrEP users with good adherence).

Exclusion Criteria:

* Have a serious cognitive or psychiatric problem that would compromise ability to provide informed consent
* Have active suicidal ideation or major mental illness (e.g., untreated psychosis or mania) at the time of interview (patients will be referred for treatment)
* Laboratory or clinical findings that would preclude PrEP initiation (e.g., decreased creatinine clearance)

Healthcare providers

Inclusion Criteria:

* Have at least 1-year experience working with HIV-negative transgender women, including providing PrEP prescription and counseling

Exclusion Criteria:

* None

Aim 2:

Inclusion Criteria:

* Age 16-29 years old
* Male sex at birth
* Self-identifies as woman or transgender women or culturally identifies with the female spectrum
* Confirmed HIV-negative status
* Self-reported recent history of condomless sex in the past 6 months
* Able to understand, read and speak Thai
* Either having not started PrEP (Group 1: PrEP naive), currently on PrEP but not adherent to PrEP (taking ≤3 pills/week) in the past month (Group 2: PrEP users).

Exclusion Criteria:

* Have a serious cognitive or psychiatric problem that would compromise ability to provide informed consent
* Have active suicidal ideation or major mental illness (e.g., untreated psychosis or mania) at the time of interview (patients will be referred for treatment)
* Laboratory or clinical findings that would preclude PrEP initiation (e.g., decreased creatinine clearance)
* Currently enrolled in another HIV intervention study

Ages: 16 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Transgender Women
Enrollment: 145 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability: System Usability Score | Month 3
  System Usability Score (SUS) is a 10-item, Likert scale used to calculate intervention usability. Each item ranges from 0 to 4 (with 4 being the most positive response). For odd-numbered items, the score is calculated by subtracting one from the user response. For even-numbered items, the score is calculated by subtracting the user response from 5. Then sum the total score and multiply that by 2.5. The overall SUS scores range from 0 to 100. A score of > 50 indicates that the technology-based interventions are acceptable.
Intervention Acceptability: System Usability Score | Month 6
  System Usability Score (SUS) is a 10-item, Likert scale used to calculate intervention usability. Each item ranges from 0 to 4 (with 4 being the most positive response). For odd-numbered items, the score is calculated by subtracting one from the user response. For even-numbered items, the score is calculated by subtracting the user response from 5. Then sum the total score and multiply that by 2.5. The overall SUS scores range from 0 to 100. A score of > 50 indicates that the technology-based interventions are acceptable.
Intervention Acceptability: Client Satisfaction Questionnaire | Month 3
  Client Satisfaction Questionnaire (CSQ-8) is an 8-items, Likert scale measuring the construct of global intervention satisfaction. The total possible composite score range from 8 to 32, with higher scores indicating a greater degree of acceptability.
Intervention Acceptability: Client Satisfaction Questionnaire | Month 6
  Client Satisfaction Questionnaire (CSQ-8) is an 8-items, Likert scale measuring the construct of global intervention satisfaction. The total possible composite score range from 8 to 32, with higher scores indicating a greater degree of acceptability.
Intervention Acceptability: Exit Interview | Month 1
  Intervention acceptability will be assess by the number of positive responses based on the exit interviews administered at month 1. Participants will be asked to provide feedback on experiences using MES-PrEP and enhanced YaCool, acceptability and ease of use, suggestions for improvement, role in PrEP uptake and adherence, and interest in continued intervention use, as well as experiences following a PrEP regimen, reasons for discontinuation of PrEP, and additional tools that would assist them in taking PrEP.
Intervention Feasibility: Number of responses to text messages | Baseline through Month 12
  Intervention feasibility will be measured by total number of responses to and frequency of usage of Enhanced YaCool. Point estimates of >50% of participants responded to Enhanced YaCool at least once is considered as the minimum criteria for feasibility.
Intervention Feasibility: Number of intervention sessions completed | Baseline through Month 12
  Intervention feasibility will be measured by number of intervention sessions completed. Point estimates of >50% of participants completed at least one intervention session is considered as the minimum criteria for feasibility.
Intervention Feasibility: Participant retention | Baseline through Month 6
  Intervention Feasibility will be measured by participants retention rate at Month 6. Retention rate of >85% at month 6 is considered as the minimum criteria for feasibility.
PrEP Adherence: Visual analog scale | Baseline through Month 12
  PrEP adherence will be measured from Young Adult Adherence Interview via computer-assisted self-interview (CASI) survey which contains a visual analog scale (VAS). VAS ranges from 0 to 100, with higher percentage indicating greater adherence to PrEP.
PrEP Adherence: Self-reported adherence | Baseline through Month 12
  PrEP adherence will be measured from self-reported adherence to PrEP in the past 4 weeks via CASI survey. The scale ranges from 0 to 100%, with higher percentage indicating greater adherence to PrEP. The result of this self-reported adherence will be triangulated with the results of dried blood spots testing.
PrEP Adherence: Dried blood spots | Baseline through Month 12
  PrEP adherence will be measured by the level of tenofovir in dried blood spots (DBS). DBS report on 80% Truvada adherence after at least three weeks of regular adherence.
PrEP Uptake | Month 1 through Month 12
  PrEP uptake will be measured by the number of PrEP prescription, using a self-report measure (participants reporting if they left the clinic with PrEP) and confirming with clinic records.

SECONDARY OUTCOMES:
PrEP Knowledge | Baseline to Month 12
  Knowledge of PrEP will be measured using the 13-item PrEP knowledge scale. The total possible score is 13, with higher scores indicating a greater degree of PrEP knowledge.
HIV Knowledge | Baseline to Month 12
  Knowledge of HIV transmission risk will be assessed using am 18-item HIV Knowledge Questionnaire. The total possible composite score range from 0 to 18, with higher scores indicating a greater degree of HIV knowledge.
Motivation: Rollnick's Readiness Ruler | Baseline to Month 12
  Behavioral intentions will be measured using 5-item Rollnick's Readiness Ruler, which correspond to PrEP uptake and adherence. Each item ranges from 0 to 10, with higher numbers indicate greater readiness for change.
Motivation: Decisional Balance for PrEP Use | Baseline to Month 12
  Attitude towards PrEP will be measured using 36-item Decisional Balance for PrEP Use. The 5-point Likert scale assesses the pros and cons of PrEP use and is helpful in understanding cognitive and motivational aspects of decision making.
Behavior skills | Baseline to Month 12
  Behavior skills will be assessed using the 8-item adapted version of Self-Efficacy for Health Promotion and Risk Reduction Questionnaire. The 5-point Likert scale assesses the confidence in using a condom, taking PrEP as recommended and getting PrEP refills. The total possible score is 40, with higher scores indicating a greater confidence for each item.
HIV Status | Baseline to Month 12
  HIV status based on 4th generation HIV-1/2 antigen/antibody combo testing.
Sexually Transmitted Infections (STIs) Diagnosis | Baseline to Month 12
  STI diagnosis based on treponemal test with rapid plasma reagin (RPR) confirmation for syphilis. Pooled urine, oropharyngeal and rectal swabs for gonorrhea and chlamydia nucleic acid amplification test (NAAT) testing.
Sexual Risk | Baseline to Month 12
  Sexual risk will be assessed through Timeline Followback via CASI, which collects sexual behavior in the past 30 days, including questions about condom use and number of sexual partners.

OTHER OUTCOMES:
Drug/Alcohol Use: ASSIST | Baseline to Month 12
  Drug/Alcohol Use will be assessed using Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) developed by the World Health Organization (WHO). ASSIST is a questionnaire that is used for identification of substance use related health risks and substance use disorders. Each item ranges from 0-12, with 0 reflecting low risk score. The total possible score is 24, with higher number indicating higher risk of health and other problems based from the current pattern of substance use.
Drug/Alcohol Use: AUDIT-C | Baseline to Month 12
  Alcohol Use Disorders Identification Test (AUDIT-C) or a brief alcohol screening instrument will also be used to identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). Each item ranges from 0 to 4, with 0 reflecting no alcohol use. The total possible score is 12, with higher number indicating higher drink above recommended limits and are at increased risks for harm.
Mental Health | Baseline to Month 12
  Mental Health will be assessed using the 12-item Thai General Health Questionnaire. The 4-point Likert scale measures psychological distress such as depression, anxiety, social impartment and somatic complaints. The total possible score is 48, with higher scores indicating higher severity of psychological distress.
Perceived HIV risk | Baseline to Month 12
  Perceived HIV risk will be measured using the 8-item Perceived Risk of HIV Scale. All items are rated on a 4-point Likert scale. The total possible score is 40, with higher scores indicating higher perception of HIV risk.
Social support | Baseline to Month 12
  Social support will be assessed using the 13-item Social Provision Scale (SPS). The 5-point Likert scale measures the availability of social support, including emotional support, information support, instrumental support, companionship and social isolation. The total possible score is 65, with higher scores indicating greater availability of social support.
PrEP stigma | Baseline to Month 12
  PrEP-related stigma will be assessed using the 10-item PrEP stigma and positive attitudes scale. The 5-point Likert scale measures opinions about PrEP. Higher scores indicate higher perceived stigma related to PrEP.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, Principal Investigator — University of Massachusetts, Worcester
Locations (3):
- Thailand (3):
  - Rainbow Sky Association of Thailand, Bangkok, Bangkok
  - Institute of HIV Research and Innovation, Bangkok, Bangkok
  - SWING Foundation, Bangkok, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wises to access the data.

REFERENCES:
- [Background] Baral SD, Poteat T, Stromdahl S, Wirtz AL, Guadamuz TE, Beyrer C. Worldwide burden of HIV in transgender women: a systematic review and meta-analysis. Lancet Infect Dis. 2013 Mar;13(3):214-22. doi: 10.1016/S1473-3099(12)70315-8. Epub 2012 Dec 21. PMID 23260128
- [Background] Logie CH, Newman PA, Weaver J, Roungkraphon S, Tepjan S. HIV-Related Stigma and HIV Prevention Uptake Among Young Men Who Have Sex with Men and Transgender Women in Thailand. AIDS Patient Care STDS. 2016 Feb;30(2):92-100. doi: 10.1089/apc.2015.0197. Epub 2016 Jan 20. PMID 26788978
- [Background] Ramautarsing RA, Meksena R, Sungsing T, Chinbunchorn T, Sangprasert T, Fungfoosri O, Meekrua D, Sumalu S, Pasansai T, Bunainso W, Wongsri T, Mainoy N, Colby D, Avery M, Mills S, Vannakit R, Phanuphak P, Phanuphak N. Evaluation of a pre-exposure prophylaxis programme for men who have sex with men and transgender women in Thailand: learning through the HIV prevention cascade lens. J Int AIDS Soc. 2020 Jun;23 Suppl 3(Suppl 3):e25540. doi: 10.1002/jia2.25540. PMID 32602660
- [Background] Rael CT, Martinez M, Giguere R, Bockting W, MacCrate C, Mellman W, Valente P, Greene GJ, Sherman S, Footer KHA, D'Aquila RT, Carballo-Dieguez A. Barriers and Facilitators to Oral PrEP Use Among Transgender Women in New York City. AIDS Behav. 2018 Nov;22(11):3627-3636. doi: 10.1007/s10461-018-2102-9. PMID 29589137
- [Background] Wood S, Gross R, Shea JA, Bauermeister JA, Franklin J, Petsis D, Swyryn M, Lalley-Chareczko L, Koenig HC, Dowshen N. Barriers and Facilitators of PrEP Adherence for Young Men and Transgender Women of Color. AIDS Behav. 2019 Oct;23(10):2719-2729. doi: 10.1007/s10461-019-02502-y. PMID 30993479
- [Background] Fuchs JD, Stojanovski K, Vittinghoff E, McMahan VM, Hosek SG, Amico KR, Kouyate A, Gilmore HJ, Buchbinder SP, Lester RT, Grant RM, Liu AY. A Mobile Health Strategy to Support Adherence to Antiretroviral Preexposure Prophylaxis. AIDS Patient Care STDS. 2018 Mar;32(3):104-111. doi: 10.1089/apc.2017.0255. PMID 29565183
- [Background] Songtaweesin WN, Kawichai S, Phanuphak N, Cressey TR, Wongharn P, Saisaengjan C, Chinbunchorn T, Janyam S, Linjongrat D, Puthanakit T; CE-PID - TRC Adolescent Study Team. Youth-friendly services and a mobile phone application to promote adherence to pre-exposure prophylaxis among adolescent men who have sex with men and transgender women at-risk for HIV in Thailand: a randomized control trial. J Int AIDS Soc. 2020 Sep;23 Suppl 5(Suppl 5):e25564. doi: 10.1002/jia2.25564. PMID 32869511
- [Background] Naar-King S, Parsons JT, Johnson AM. Motivational interviewing targeting risk reduction for people with HIV: a systematic review. Curr HIV/AIDS Rep. 2012 Dec;9(4):335-43. doi: 10.1007/s11904-012-0132-x. PMID 22890780
- [Background] Bonar EE, Wolfe JR, Drab R, Stephenson R, Sullivan PS, Chavanduka T, Hailu B, Guest JL, Bauermeister J. Training Young Adult Peers in a Mobile Motivational Interviewing-Based Mentoring Approach to Upstream HIV Prevention. Am J Community Psychol. 2021 Mar;67(1-2):237-248. doi: 10.1002/ajcp.12471. Epub 2020 Nov 2. PMID 33137221
- [Background] Dale SK. Using Motivational Interviewing to Increase PrEP Uptake Among Black Women at Risk for HIV: an Open Pilot Trial of MI-PrEP. J Racial Ethn Health Disparities. 2020 Oct;7(5):913-927. doi: 10.1007/s40615-020-00715-9. Epub 2020 Feb 20. PMID 32078743
- [Background] Naar-King S, Outlaw AY, Sarr M, Parsons JT, Belzer M, Macdonell K, Tanney M, Ondersma SJ; Adolescent Medicine Network for HIV/AIDS Interventions. Motivational Enhancement System for Adherence (MESA): pilot randomized trial of a brief computer-delivered prevention intervention for youth initiating antiretroviral treatment. J Pediatr Psychol. 2013 Jul;38(6):638-48. doi: 10.1093/jpepsy/jss132. Epub 2013 Jan 28. PMID 23359664
- [Background] Dubov A, Altice FL, Fraenkel L. An Information-Motivation-Behavioral Skills Model of PrEP Uptake. AIDS Behav. 2018 Nov;22(11):3603-3616. doi: 10.1007/s10461-018-2095-4. PMID 29557540
- [Background] Phanuphak N, Anand T, Jantarapakde J, Nitpolprasert C, Himmad K, Sungsing T, Trachunthong D, Phomthong S, Phoseeta P, Tongmuang S, Mingkwanrungruang P, Meekrua D, Sukthongsa S, Hongwiangchan S, Upanun N, Barisri J, Pankam T, Phanuphak P. What would you choose: Online or Offline or Mixed services? Feasibility of online HIV counselling and testing among Thai men who have sex with men and transgender women and factors associated with service uptake. J Int AIDS Soc. 2018 Jul;21 Suppl 5(Suppl Suppl 5):e25118. doi: 10.1002/jia2.25118. PMID 30033644
- [Background] Janamnuaysook R, Guo Y, Yu YJ, Phanuphak N, Kawichai S, MacDonell K, Jupimai T, Rongkavilit C, Wang B. Lived experiences with pre-exposure prophylaxis uptake and adherence among transgender women in Thailand: a qualitative study. Sex Health. 2024 Jan;21:SH23102. doi: 10.1071/SH23102. PMID 38219741
- [Derived] MacDonell KK, Wang B, Phanuphak N, Janamnuaysook R, Srimanus P, Rongkavilit C, Naar S. Optimizing an mHealth Intervention to Improve Uptake and Adherence to HIV Pre-exposure Prophylaxis in Young Transgender Women: Protocol for a Multi-Phase Trial. JMIR Res Protoc. 2022 May 19;11(5):e37659. doi: 10.2196/37659. PMID 35587370